CLINICAL TRIAL: NCT03980249
Title: A Pilot Study: Evaluating the Anti-Cancer Effects of Carvedilol With TTFields and Standard of Care in Glioblastoma and Response of Peripheral Glioma Circulating Tumor Cells
Brief Title: Anti-Cancer Effects of Carvedilol With Standard Treatment in Glioblastoma and Response of Peripheral Glioma Circulating Tumor Cells
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: West Virginia University (Other)
Collaborators: NovoCure Ltd. (Industry); West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU020318
Record Dates: First submitted 2019-05-01; First posted 2019-06-10 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Carvedilol + Standard Treatment (Experimental): Subjects will receive carvedilol starting at 6.25 mg orally (PO) twice daily for 1-2 weeks and if tolerated will then be increased to 12.5 mg PO twice daily starting on day 1 of concurrent chemoradiotherapy and continue daily until the end of adjuvant cycle 6 of temozolomide and Tumor Treated Fields.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol: Start at 6.26 mg PO twice daily for 1-2 weeks and if tolerated, will be increased to 12.5 mg PO twice daily for 6 cycles as tolerated.
  Other Names: Coreg

SUMMARY:
The purpose of this pilot study is to evaluate the addition of carvedilol with standard of care treatment to determine if it will improve progression-free survival in the front line setting in patients with glioblastoma multiforme (GBM). In addition, monitoring of circulating tumor cells (CTCs) by a real-time reverse transcriptase polymerase chain reaction (qRT-PCR) assay to correlate with the clinical findings.

DETAILED DESCRIPTION:
This is a pilot study to assess efficacy of the addition of a non-selective beta-blocker to standard of care treatment in the front-line setting of glioblastoma multiforme. And to also evaluate the level of peripheral glioma circulating tumor cells via TeleomeScan assay to correlate disease response determined by neuro-imaging.

Peripheral blood samples will be collected at baseline, on day 1 of cycle 1 and then after on day 1 of cycle 4 and at the end of cycle 6 of adjuvant chemotherapy. in order to correlate the biological effects of treatment response. The investigators will evaluate the quantity of peripheral glioma circulating tumor cells and want to apply the information seen in the periphery to the status of the cancer on imaging studies.

Subjects will start oral carvedilol at 6.25 mg orally twice daily and will evaluate the patient and vital status if they tolerate this dose at 1-2 weeks after initiation. If tolerated well, will increase the dose to the maximum anticipation of 12.5 mg orally twice daily. Treatment will proceed for 6 cycles and carvedilol will stop at the end of 6 cycles. Patients will be monitored with neuroimaging prior before chemoradiotherapy, before adjuvant temozolomide and every 2 months on adjuvant temozolomide. Following the completion of 6 cycles of adjuvant therapy, patients will continue to receive neuroimaging on every 3 months' basis until disease progression based upon standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed WHO Grade IV Glioblastoma
* Subjects must have not received previous chemotherapy or radiation therapy for GBM
* Subjects must have systolic blood pressure greater than or equal to 90 and heart rate >59
* Subjects who are on beta-blockers for other etiologies may enroll on study and switch therapy to carvedilol if deemed medical appropriate per treating physician

Exclusion Criteria:

* Subjects receiving any other investigational agents
* Subjects who have severe and uncontrolled asthma, COPD
* Systolic blood pressure <90 mmHg or HR <60 bpm without antihypertensive medications at baseline
* Subjects with uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Allergy to beta blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Survival curve of overall survival | From start of carvedilol treatment until the date of first documented progression or death which ever comes first (approximately 6-15 months)
  Kaplan-Meier curves for overall survival in order to see if the addition of carvedilol to standard of care appears promising from a clinical standpoint
Survival curve of progression free survival | From start of carvedilol treatment until the date of first documented progression or death which ever comes first (approximately 6-15 months)
  Kaplan-Meier curves for progression free survival in order to see if the addition of carvedilol to standard of care appears promising from a clinical standpoint

SECONDARY OUTCOMES:
Quantify Circulating Tumor Cells (CTCs) | Baseline (prior to any treatment), Cycle 1 Day 1, Cycle 4 day 1, End of cycle 6 of Chemotherapy (each cycle is 28 days)
  Quantify CTCs via qRT-PCR assay and to assess how the trend of CTCs correspond to disease status as measured by RANO criteria on neuro-imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kolodney, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Cancer Institute - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03980249/ICF_000.pdf